CLINICAL TRIAL: NCT07036302
Title: Clinical Evaluation of Trichloroacetic Chemical Peel And Fractional Laser: Comparative Analysis Of Quantitative And Qualitative Parameters
Brief Title: Comparative Effects Of Trichloroacetic Chemical Peel And Fractional Laser
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Roberto Cortelli (Other)
Collaborators: Cavalca & Cortelli private research center (Unknown)
Responsible Party: Sponsor-Investigator, Jose Roberto Cortelli, Professor and Doctorate, University of Taubate
Organization: University of Taubate (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 84943324.1.0000.5501
Record Dates: First submitted 2025-06-15; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Melasma; Acne Scars - Mixed Atrophic and Hypertrophic; Resurfacing; Rejuvenation
Keywords: chemical peel; Er-YAG; ND-YAG; fractional laser; home care
MeSH Terms: conditions — Melanosis; Hypertrophy | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistics staff
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Melasma TCA associated with croton oil peel (Experimental): 3 sections every 30 days of a chemical peel combining 35% TCA and croton oil in the same formulation
  Interventions: Procedure: 35% TCA combined with croton oil peel
- Melasma isolate TCA peel (Active Comparator): 3 sections every 30 days of a chemical peel containing only 35% TCA
  Interventions: Procedure: Isolate 35% TCA peel
- Melasma Laser ND-YAG laser (Active Comparator): 3 sections every 30 days of Neodymium: yttrium-aluminum-garnet (ND-YAG) laser
  Interventions: Radiation: Neodymium -YAG laser Q-switched
- Acne scars TCA associated with croton oil peel (Experimental): 3 sections every 30 days of a chemical peel combining 35% TCA and croton oil in the same formulation
  Interventions: Procedure: 35% TCA combined with croton oil peel
- Acne scars isolate TCA peel (Active Comparator): 3 sections every 30 days of a chemical peel containing only 35% TCA
  Interventions: Procedure: Isolate 35% TCA peel
- Acne scars Er-YAG laser (Active Comparator): 3 sections every 30 days of Erbium: yttrium-aluminum-garnet (Er-YAG) laser
  Interventions: Radiation: Erbium-YAG laser
- Facial rejuvenation TCA associated with croton oil peel (Experimental): 3 sections every 30 days of a chemical peel combining 35% TCA and croton oil in the same formulation
  Interventions: Procedure: 35% TCA combined with croton oil peel
- Facial rejuvenation isolate 35% TCA peel (Active Comparator): 3 sections every 30 days of a chemical peel containing only 35% TCA
  Interventions: Procedure: Isolate 35% TCA peel
- Facial wrinkles Er-YAG laser (Active Comparator): 3 sections every 30 days of Erbium: yttrium-aluminum-garnet (Er-YAG) laser
  Interventions: Radiation: Erbium-YAG laser

INTERVENTIONS:
Procedure: 35% TCA combined with croton oil peel — 3 sections every 30 days of 35% TCA combined with croton oil peel
  Arms: Acne scars TCA associated with croton oil peel; Facial rejuvenation TCA associated with croton oil peel; Melasma TCA associated with croton oil peel
Procedure: Isolate 35% TCA peel — 3 sections every 30 days of isolate 35% TCA peel
  Arms: Acne scars isolate TCA peel; Facial rejuvenation isolate 35% TCA peel; Melasma isolate TCA peel
Radiation: Erbium-YAG laser — 3 sections every 30 days of Er-YAG laser
  Arms: Acne scars Er-YAG laser; Facial wrinkles Er-YAG laser
Radiation: Neodymium -YAG laser Q-switched — 3 sections every 30 days of ND-YAG laser
  Arms: Melasma Laser ND-YAG laser

SUMMARY:
More than aesthetics, the search for orofacial harmonization treatments has increased when the negative emotional impact of some facial conditions such as melasma and acne scars is recognized. This study will evaluate the effects of chemical peels with 35% TCA (trichloroacetic acid) and two types of fractional laser in orofacial harmonization procedures. A sample of 100-120 participants at least 18 years of age, male or female, with complaints of melasma (n=36 to 40), acne scars (n=36 to 40) or facial wrinkles (n=36 to 40) will be recruited to underwent 3 consecutive treatment sections every 30 days. Besides clinical improvements, global satisfaction scale of the professional and the patient will be measured in addition to the impact of the treatment on the quality of life of the participants and the sensory experience in relation to pain. Pre- and pos-peeling home care will be provided to measure whether they influence results or not. The aim of this study is to identify the most appropriate treatment strategy for frequent complaints in clinical practice, and among them, the one that promotes the best experience, with the shortest recovery time and is cost-effective.

DETAILED DESCRIPTION:
More than aesthetics, the search for orofacial harmonization treatments has increased when the negative emotional impact of some facial conditions such as melasma and acne scars is recognized. This randomized clinical trial will evaluate the effects of chemical peel with 35% TCA (trichloroacetic acid)associated with croton oil. And to compare the results with its isolated formulation containing only 35% TCA and with two types of fractional laser (2940nm Er-YAG and 1640nm Nd-YAG) in orofacial harmonization procedures. This study will be based on a sample of 100-120 participants at least 18 years of age, male or female, with complaints of melasma (n=36 to 40), acne scars (n=36 to 40) or facial wrinkles (n=36 to 40). The experimental times will be day -15 (pre-treatment), day 0 (1st treatment session), day 30 (2nd treatment session), day 60 (3rd treatment session), day 70 (immediate post-treatment) and day 120 (mediate post-treatment). The primary outcomes will be the difference (pre- versus post-peeling) in the scores of Melasma (mMASI), acne scars (SCAR-S) or facial wrinkles (Glogau index), in the respective groups according to the main complaints. As secondary outcomes, the global satisfaction scale of the professional (PGA) and the patient (PtGA) will be measured; the impact of the treatment on the quality of life of the participants (SKINDEX-16) and the sensory experience in relation to pain (EVA 1 to 10). All participants, under local anesthesia (button anesthesia), will be randomized into one of three treatment groups: 35% TCA associated with croton oil (test), 35% TCA alone, Er-Yag or Nd-YAG laser (comparators). Intra- and inter-group differences will be considered statistically significant when p < 0.05. The aim of this study is to identify the most appropriate treatment strategy for frequent complaints in clinical practice, and among them, the one that promotes the best experience, with the shortest recovery time and is cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* aged 18 or over
* acne scars, melasma or clear signs of photoaging and evident wrinkles
* participants with acne scars or melasma will be included if they have never undergone treatment or if previous treatment has been ineffective.

Exclusion Criteria:

* phototype VI
* autoimmune and dermatological diseases
* known allergies to the components of the formulations
* patients who prefer other treatment options
* history of keloids
* pregnant women
* breastfeeding women
* women of childbearing age who do not adopt a valid method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glogau scale | Baseline versus 3 months
  Changes in Glogau scale (I to IV) for rejuvenation group. Higher values indicate worse aging conditions.
Melasma index | baseline versus 3 months after treatment
  Changes in 1 to 6 scores of modified Melasma Area and Severity Index (mMASI). Higher values indicate worse melasma conditions.
Acne Scars Index | Baseline versus 3 months after treatment
  Changes in Global 1 to 5 Scale for Acne Scar Severity (SCAR-S). Higher values indicate worse acne scars conditions.

SECONDARY OUTCOMES:
Treatment impact on Quality of life | Baseline versus immediate post-treatment
  SKINDEX-16 scores (0 to 100) after treatment. Higher values indicate worse quality of life.
Patient's satisfaction | Immediate post-treatment
  Evaluation of Patient Global Assessment (PtGA) instrument. Results are expressed into quartile percentages. The most higher percentages indicates the best patient's satisfaction.
Professional's satisfaction | 3 months after treatment
  Evaluation of Physician Global Assessment (PGA) instrument. Results are expressed into quartile percentages. The most higher percentages indicates the best professional's satisfaction.

OTHER OUTCOMES:
Self-reported pain | Days 0, 30 and 60.
  Evaluation by a 10 point Visual Analogue Scale. Higher values indicate worse pain experience.
Adverse Events | Baseline versus 12 months after treatment
  Self-reported and diagnosed adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sheila C Cortelli, Doctorate, Principal Investigator — University of Taubate
Locations (2):
- Brazil (2):
  - Cavalca & Cortelli Research Center, Taubaté, São Paulo
  - University of Taubate Dental School, Taubaté, São Paulo

IPD SHARING:
Plan to Share IPD: No
Only not identified data will be shared within research team.